CLINICAL TRIAL: NCT07057102
Title: Applications of Multiple Omics Sequencing Technologies in Predicting the Efficacy and Monitoring the Recurrence of Non-Small Cell Lung Cancer: A Prospective, Non-Interventional Study
Brief Title: Multiple Omics Sequencing Technologies in Predicting the Efficacy and Monitoring the Recurrence of Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhijie Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC5160
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; ctDNA; MRD
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Advanced/Metastatic: Advanced/Metastatic non-small cell lung cancer
- Neoadjuvant Therapy: Non-small cell lung cancer patients undergoing neoadjuvant therapy
- Adjuvant therapy: Non-small cell lung cancer patients undergoing adjuvant therapy after surgery

SUMMARY:
Lung cancer is one of the diseases with the highest global incidence and mortality. Studies have confirmed that liquid biopsy markers such as minimal residual disease (MRD) detection in solid tumors, circulating tumor DNA (ctDNA), and T-cell receptor (TCR) have roles in monitoring disease status, prognostic evaluation, recurrence prediction, and guiding treatment decisions in NSCLC patients. Peripheral blood dynamic monitoring indicators have broad application prospects and may completely transform the treatment paradigm for NSCLC patients in the future. However, current limitations exist, including the need to improve the sensitivity of detection methods, the lack of uniform criteria for defining MRD positivity, the undetermined timing and cycle of MRD testing, and insufficient results from large-scale prospective clinical trials. Therefore, the transition of peripheral blood-based dynamic testing to routine clinical practice still requires results from large-scale prospective clinical trials. This study intends to conduct a prospective clinical trial enrolling NSCLC patients with different stages and treatment modalities (immunotherapy combined with chemotherapy, targeted therapy combined with chemotherapy, neoadjuvant therapy, adjuvant therapy). Based on peripheral blood and tumor tissue samples, it will systematically integrate multi-omics approaches including ctDNA testing, whole exome sequencing (WES), genome-wide methylation sequencing (GM-seq), and TCR-seq to carry out comprehensive, precise, and dynamic biomarker detection for efficacy monitoring and recurrence prediction, providing new methods and evidence for the clinical application of dynamic liquid biopsy monitoring in lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent;
2. Aged 18 years or older;
3. Expected life expectancy of ≥3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 (see Appendix 1);
5. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) patients;
6. Classified as stage II, III, or IV according to the AJCC TNM staging system (9th edition);
7. Willing to provide blood samples and pre-treatment paraffin-embedded tissue samples;
8. With evaluable target lesions for efficacy assessment.

Exclusion Criteria

1. In the investigator's opinion, unsuitable for peripheral blood collection due to complications or other circumstances;
2. Active, known, or suspected autoimmune diseases (except vitiligo, type 1 diabetes, residual hypothyroidism caused by autoimmune thyroiditis requiring only hormone replacement therapy, or conditions not expected to relapse without external stimulation);
3. Active tuberculosis (TB) infection confirmed by chest X-ray, sputum examination, and clinical physical examination. Patients with a history of active TB infection within the past 1 year, even if treated, will be excluded. Patients with a history of active TB infection more than 1 year ago will also be excluded unless they can demonstrate that previous antitubercular treatment was fully effective;
4. Comorbidities requiring treatment with immunosuppressive drugs, or comorbidities requiring systemic or local corticosteroids at immunosuppressive doses;
5. Pregnant or lactating;
6. Positive for human immunodeficiency virus antibody (HIVAb), active hepatitis B virus infection (HBsAg-positive and HBV-DNA > 10³ copies/ml), or hepatitis C virus infection (HCV antibody-positive and HCV-RNA > the lower limit of detection at the study center);
7. History of severe neurological or psychiatric disorders, including but not limited to: dementia, depression, seizures, bipolar disorder, etc.;
8. Use of any antitumor-active drugs prior to blood sample collection;
9. Previous history of other malignancies (excluding non-melanoma skin cancer and the following in situ carcinomas: bladder, stomach, colon, endometrium, cervix/dysplasia, melanoma, or breast cancer);
10. Administration of live vaccines within 28 days prior to blood sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients From Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Liquid Biopsy Biomarkers | From enrollment to the end of monitoring at 3 years or the occurrence of disease progression.
  Liquid biopsy biomarkers for efficacy monitoring, prognostic evaluation, and recurrence prediction

SECONDARY OUTCOMES:
Comparison of MRD and Conventional Imaging | From enrollment to the end of monitoring at 3 years or the occurrence of disease progression.
  Compare the efficacy of minimal residual disease (MRD) and conventional imaging in monitoring disease status, prognostic evaluation, and recurrence prediction.
The appropriate timing for minimal residual disease (MRD) testing | From enrollment to the end of monitoring at 3 years or the occurrence of disease progression.
  To explore the appropriate timing for minimal residual disease (MRD) testing during the diagnosis and treatment process of NSCLC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijie Wang, MD, Study Director — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellini B, Chaudhuri AA. Circulating Tumor DNA Minimal Residual Disease Detection of Non-Small-Cell Lung Cancer Treated With Curative Intent. J Clin Oncol. 2022 Feb 20;40(6):567-575. doi: 10.1200/JCO.21.01929. Epub 2022 Jan 5. PMID 34985936
- [Background] Fujimoto D, Yoshioka H, Kataoka Y, Morimoto T, Hata T, Kim YH, Tomii K, Ishida T, Hirabayashi M, Hara S, Ishitoko M, Fukuda Y, Hwang MH, Sakai N, Fukui M, Nakaji H, Morita M, Mio T, Yasuda T, Sugita T, Hirai T. Pseudoprogression in Previously Treated Patients with Non-Small Cell Lung Cancer Who Received Nivolumab Monotherapy. J Thorac Oncol. 2019 Mar;14(3):468-474. doi: 10.1016/j.jtho.2018.10.167. Epub 2018 Nov 20. PMID 30468872
- [Background] Dong S, Wang Z, Zhang JT, Yan B, Zhang C, Gao X, Sun H, Li YS, Yan HH, Tu HY, Liu SM, Gong Y, Gao W, Huang J, Liao RQ, Lin JT, Ke EE, Xu Z, Zhang X, Xia X, Li AN, Liu SY, Pan Y, Yang JJ, Zhong WZ, Yi X, Zhou Q, Yang XN, Wu YL. Circulating Tumor DNA-Guided De-Escalation Targeted Therapy for Advanced Non-Small Cell Lung Cancer: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Jul 1;10(7):932-940. doi: 10.1001/jamaoncol.2024.1779. PMID 38869865
- [Background] Mack PC, Miao J, Redman MW, Moon J, Goldberg SB, Herbst RS, Melnick MA, Walther Z, Hirsch FR, Politi K, Kelly K, Gandara DR. Circulating Tumor DNA Kinetics Predict Progression-Free and Overall Survival in EGFR TKI-Treated Patients with EGFR-Mutant NSCLC (SWOG S1403). Clin Cancer Res. 2022 Sep 1;28(17):3752-3760. doi: 10.1158/1078-0432.CCR-22-0741. PMID 35713632
- [Background] Hellmann MD, Nabet BY, Rizvi H, Chaudhuri AA, Wells DK, Dunphy MPS, Chabon JJ, Liu CL, Hui AB, Arbour KC, Luo J, Preeshagul IR, Moding EJ, Almanza D, Bonilla RF, Sauter JL, Choi H, Tenet M, Abu-Akeel M, Plodkowski AJ, Perez Johnston R, Yoo CH, Ko RB, Stehr H, Gojenola L, Wakelee HA, Padda SK, Neal JW, Chaft JE, Kris MG, Rudin CM, Merghoub T, Li BT, Alizadeh AA, Diehn M. Circulating Tumor DNA Analysis to Assess Risk of Progression after Long-term Response to PD-(L)1 Blockade in NSCLC. Clin Cancer Res. 2020 Jun 15;26(12):2849-2858. doi: 10.1158/1078-0432.CCR-19-3418. Epub 2020 Feb 11. PMID 32046999
- [Background] Provencio M, Serna-Blasco R, Nadal E, Insa A, Garcia-Campelo MR, Casal Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Calvo V, Martin-Lopez J, Garcia-Garcia F, Casarrubios M, Franco F, Sanchez-Herrero E, Massuti B, Cruz-Bermudez A, Romero A. Overall Survival and Biomarker Analysis of Neoadjuvant Nivolumab Plus Chemotherapy in Operable Stage IIIA Non-Small-Cell Lung Cancer (NADIM phase II trial). J Clin Oncol. 2022 Sep 1;40(25):2924-2933. doi: 10.1200/JCO.21.02660. Epub 2022 May 16. PMID 35576508
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- [Background] Gale D, Heider K, Ruiz-Valdepenas A, Hackinger S, Perry M, Marsico G, Rundell V, Wulff J, Sharma G, Knock H, Castedo J, Cooper W, Zhao H, Smith CG, Garg S, Anand S, Howarth K, Gilligan D, Harden SV, Rassl DM, Rintoul RC, Rosenfeld N. Residual ctDNA after treatment predicts early relapse in patients with early-stage non-small cell lung cancer. Ann Oncol. 2022 May;33(5):500-510. doi: 10.1016/j.annonc.2022.02.007. Epub 2022 Mar 17. PMID 35306155
- [Background] Zhang JT, Liu SY, Gao W, Liu SM, Yan HH, Ji L, Chen Y, Gong Y, Lu HL, Lin JT, Yin K, Jiang BY, Nie Q, Liao RQ, Dong S, Guan Y, Dai P, Zhang XC, Yang JJ, Tu HY, Xia X, Yi X, Zhou Q, Zhong WZ, Yang XN, Wu YL. Longitudinal Undetectable Molecular Residual Disease Defines Potentially Cured Population in Localized Non-Small Cell Lung Cancer. Cancer Discov. 2022 Jul 6;12(7):1690-1701. doi: 10.1158/2159-8290.CD-21-1486. PMID 35543554
- [Background] Chaudhuri AA, Chabon JJ, Lovejoy AF, Newman AM, Stehr H, Azad TD, Khodadoust MS, Esfahani MS, Liu CL, Zhou L, Scherer F, Kurtz DM, Say C, Carter JN, Merriott DJ, Dudley JC, Binkley MS, Modlin L, Padda SK, Gensheimer MF, West RB, Shrager JB, Neal JW, Wakelee HA, Loo BW Jr, Alizadeh AA, Diehn M. Early Detection of Molecular Residual Disease in Localized Lung Cancer by Circulating Tumor DNA Profiling. Cancer Discov. 2017 Dec;7(12):1394-1403. doi: 10.1158/2159-8290.CD-17-0716. Epub 2017 Sep 24. PMID 28899864
- [Background] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338